CLINICAL TRIAL: NCT07141030
Title: To Assess the Pharmacokinetic (PK) Differences of GZR18 Injection Between Subjects With Renal Impairment and Those With Normal Renal Function, Providing a Basis for Establishing a Clinical Dosing Regimen for Patients With Renal Impairment
Brief Title: Study of Pharmacokinetics and Safety of GZR18 Injection in Subjects With Renal Impairment and Normal Renal Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZR18-BWM-106
Record Dates: First submitted 2025-08-12; First posted 2025-08-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Obesity/Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GZR18 injection (Experimental)
  Interventions: Drug: GZR18 injection

INTERVENTIONS:
Drug: GZR18 injection — GZR18 injection:3mg

SUMMARY:
This study adopts a multicenter, single-dose, open-label, and parallel design, which is aimed at assessing the PK and safety profiles of GZR18 Injection in subjects with normal renal function and those with mild, moderate or severe renal impairment.

The study duration for each subject in this study is up to 50 days, including a screening period of up to 14 days (Day-14 to Day-1), an 8-day dosing/observation period (Day 1 to Day 8), and a 28-day follow-up period (Day 9 to Day 36).

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects sign the Informed Consent Form (ICF) before the study, fully understand the contents, process and possible adverse reactions of the study, and be able to follow the contraindications and restrictions specified in this protocol.

  2.Subjects (male or female) age ≥ 18 and ≤ 75 years at the time of signing ICF.

  3.Subjects with childbearing potential from signing the ICF to 8 weeks after the last dose have no family planning, are willing to adopt effective contraceptive measures and have no plans for sperm donation; women of childbearing potential are not pregnant or lactating: they must have a negative pregnancy test at screening and have no unprotected sexual intercourse within 2 weeks before screening.

  4.Subjects weighing ≥ 50 kg and 20 ≤ BMI ≤ 40 kg/m2 at screening.

  5.Subjects with normal renal function must also meet the following conditions:
  1. 90 mL/min ≤ individual's GFR < 130 mL/min at screening (see Appendix 2: Formulas Involved in the Protocol for the calculation formula).
  2. Subjects with normal laboratory test results, vital signs, ECG, physical examination, chest AP view, abdominal B-ultrasound, and other examination results at screening or without clinically significant abnormalities as assessed by the investigator.

  6.Subjects with renal impairment must also meet all of the following:
  1. Mild renal impairment group: 60 mL/min ≤ individual's GFR < 90 mL/min at screening; moderate renal impairment group: 30 mL/min ≤ individual's GFR < 60 mL/min at screening; severe renal impairment group: 15 mL/min ≤ individual's GFR < 30 mL/min at screening.
  2. Subjects with moderate and severe renal impairment should meet the diagnostic criteria for chronic kidney disease (outpatient medical records, hospitalization medical records or laboratory test results can be used as evidence). If the subject is receiving drug therapy, a stable medication regimen (at least within 2 weeks before administration) is required.

     Exclusion Criteria:
* 1.Subjects with allergic constitution, including those with a history of severe drug allergy or hypersensitivity reactions, and those known or suspected to be allergic to GLP-1 drugs or their excipients as considered by the investigator.

  2.Subjects with a history of acute or chronic pancreatitis and pancreatic injury before screening; subjects with viral hepatitis, alcoholic liver disease, hepatic cirrhosis, autoimmune hepatitis and other liver diseases before screening; subjects with symptomatic gallbladder disease at screening.

  3.Subjects who routinely receive dialysis or have a history of kidney transplantation or other organ transplantation before screening.

  4.Subjects with severe infection, severe trauma, gastrointestinal surgery, or other major surgical operations within 6 months before screening.

  5.Subjects with a history of moderate or major depression, suicidal tendency or suicidal behavior before screening; or other serious mental disorders (schizophrenia, bipolar affective disorder, etc.); or other psychiatric diseases that the investigator considers inappropriate for this study.

  6. Subjects with a history of drug abuse or drug use within 1 year before screening; or subjects with positive result in a drug abuse screening (urine) (which cannot be justified by concurrent medications, such as those used for treating pain, anxiety, or insomnia as complications of renal disorder) at screening.

  7.Subjects who have received a vaccine within 2 weeks before screening or are planning to be vaccinated during the study or within 1 month postdose.

  8.Subjects who are positive for any indicator of human immunodeficiency virus (HIV) antibody, Treponema pallidum antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or hepatitis C virus (HCV) antibody at screening.

  9.Subjects deemed unsuitable for inclusion by the investigator for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cmax:Maximum plasma concentration | through study completion, an average of 36 days
AUC0-last:Area under the plasma concentration-time curve at 0 h to last observation time-point after a single dose. | through study completion, an average of 36 days
AUC0-inf:Area under the plasma concentration-time curve at 0 h to infinity after a single dose. | through study completion, an average of 36 days

SECONDARY OUTCOMES:
AUC0-336 h：Area under the plasma concentration-time curve from time zero to 336 hours | through study completion, an average of 36 days
Tmax:Time of Maximum Drug ConcentrationTime to Maximum aentration | through study completion, an average of 36 days
TEAE：Treatment Emergent Adverse Event | through study completion, an average of 36 days

CONTACTS AND LOCATIONS:
Locations (1):
- Gan & Lee Pharmaceuticals, Beijing, China